CLINICAL TRIAL: NCT03455582
Title: Longitudinal Study of Cognition in Primary Progressive Multiple Sclerosis: a Cohort Study
Brief Title: Cognition Evolution and MRI Markers in PPMS Patients on 2 Years
Acronym: PRO-COG
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2017/14
Record Dates: First submitted 2018-01-04; First posted 2018-03-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis, Primary Progressive
Keywords: cognitive impairment; ecological assessment; brain MRI
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient (Experimental): PPMS diagnosis according to McDonald 2010 criteria (Polman et al, 2011)
  Interventions: Other: Clinical assessment; Other: Ecological evaluation; Other: Neuropsychological evaluation; Other: Psychological evaluation; Device: MRI Evaluation
- Control (Active Comparator): 40 Healthy controls
  Interventions: Other: Ecological evaluation; Other: Neuropsychological evaluation; Other: Psychological evaluation; Device: MRI Evaluation

INTERVENTIONS:
Other: Clinical assessment — Expanded Disability Status Scale (EDSS), ambulation test and Multiple Sclerosis functional composite (MSFC). Medications will be recorded.
  Arms: patient
Other: Ecological evaluation — Virtual reality task and Actual reality
Other: Neuropsychological evaluation — cognitive tests exploring information processing speed, attention/concentration, working and episodic memories and executive function
Other: Psychological evaluation — questionnaires for depression, anxiety and fatigue
Device: MRI Evaluation — morphological MRI and resting state functional MRI (fMRI)

SUMMARY:
Cognitive impairment is nowadays more and more recognized as an important feature of the multiple sclerosis (MS) disease. Cognitive disorders frequency in MS is estimated between 40 and 60%. Cognitive impairment affects quality of life and vocational status in MS patients.

Until recently, little information was available on the cognitive dysfunction and their evolution that occur in primary progressive multiple sclerosis (PPMS) as compared with relapsing-remitting MS (RRMS). In PPMS pathological studies have shown the importance of cortical demyelination and meningeal inflammation suggesting that the GM alteration could play a major role in the cognitive impairment in this phenotype. The cognitive evolution and the brain tissue alteration at the origin of these difficulties remain poorly understood in PPMS. The use of new techniques for morphological and functional MRI can study the contribution of diffuse White Matter (WM) alteration (probably through disconnexion of relevant network) and diffuse Grey matter (GM) alterations in the cerebral cortex and other structures (the hippocampi, the cerebellum, and the thalami) in cognitive impairment in PPMS patients and on their evolution.

ELIGIBILITY:
Inclusion Criteria:

PATIENTS

* Male or female;
* Age ≥ 18 years;
* PPMS diagnosis according to McDonald 2010 criteria;
* Disease duration ≤ 15 years;
* Native French speaking;
* Being affiliated to health insurance;
* Willing to participate and to sign informed consent.

HEALTHY CONTROLS

* Male or Female;
* Age ≥ 18 years;
* Native French speaking;
* Being affiliated to health insurance;
* Willing to participate and to sign informed consent.

Exclusion Criteria:

PATIENTS

* previous history of other neurological disease;
* psychiatric comorbidity including severe depression according to DSM-IV;
* alcohol or other addiction to toxic;
* disabling visual or motor problems preventing participation to neuropsychological assessments;
* change of psychotropic drug since less than one month;
* contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body,claustrophobia or refusing MRI);
* illiteracy, is unable to count or to read;
* pregnant or breastfeeding women;
* patient concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

HEALTHY CONTROLS

* history of neurological disease;
* family history of MS;
* psychiatric comorbidity including severe depression according to DSM-IV;
* alcohol or other toxic addiction;
* psychotropic drugs; known cognitive complaint or neuropsychological affection;
* prior neuropsychological testing with the same tests less than 6 months
* contra-indication to MRI (pacemakers, aneurysm clips, artificial heart valves, ear implants, meta fragments or foreign objects in the eyes, skin or body, claustrophobia or refusing MRI);
* illiteracy, is unable to count or to read;
* pregnant or breastfeeding women;
* person concerned by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change of composite z cognitive score based on individual neuropsychological scores | At baseline (day 0) and at 24 months from baseline
  The composite z cognitive score is the average of z individual cognitive scores. The score from each cognitive test is transformed into z-scores. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time (baseline and 2 years).
  Individual neuropsychological scores included in composite z cognitive score : the Alertness subtest, the divided attention subtest and the visual-scanning subtest from the TAP, The Symbol-digit-modalities-test, the Paced-Auditory-Serial-Addition-Test 3s, reversed span, the Stroop test, the Verbal fluency, Trail Making test, the California Verbal memory learning test and the Brief visual memory test -revised

SECONDARY OUTCOMES:
Correlation of composite z cognitive score and ecological score with MRI parameters reflecting grey and white matter integrity and anatomic/functional connectivity | At baseline (day 0) and at 24 months from baseline
  The composite z cognitive score is the average of z individual cognitive scores. The score from each cognitive test is transformed into z-scores. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time.
  The composite z ecological score is the average of z ecological scores of virtual reality task (Urban DailyCog©) and actual reality tests.
Change of composite z cognitive score based on individual neuropsychological scores | At baseline (day 0), at 12 months and at 24 months from baseline
  The composite z cognitive score is the average of z individual cognitive scores. The score from each cognitive test is transformed into z-scores. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time.
Changes of composite z ecological score based on individual ecological scores | At baseline (day 0), at 12 months and at 24 months from baseline
  The composite z cognitive score is the average of z individual cognitive scores. The score from each cognitive test is transformed into z-scores. Z-scores will be calculated for each cognitive score with the following formula: (patient's score - mean value of HC group matched for age, sex, and education level)/standard deviation of the matched HC for each evaluation time. The composite z ecological score is the average of z ecological scores of virtual reality task (Urban DailyCog©) and actual reality tests.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélie RUET, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - CHU de Bordeaux, Bordeaux
  - CHU de Limoges, Limoges
  - CHU de Poitiers, Poitiers